CLINICAL TRIAL: NCT00261755
Title: Acupuncture as Pain Relief and Relaxation During Childbirth. A Randomized Controlled Study
Brief Title: Acupuncture as Pain Relief and Relaxation During Childbirth
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other); Direktør E. Danielsen og Hustrus Fond (Unknown); Kong Christian den Tiendes Fond (Unknown); Lundbeck Foundation (Other); Manufacturer Mads Clausen Foundation (Other); Else og Mogens Wedell-Wedellsborgs Fond (Unknown); The Hede Nielsen Family Foundation (Other); Videns- og Forskningscenter for Alternativ Behandling (Other); DADJ (Den almindelige Danske Jordemoderforening) (Unknown)
Responsible Party: Lone Hvidman, MD,PhD, Department of Obstetrics, Aarhus University Hospital, Skejby, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Akupunktur2001-41-1305
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Acupuncture Analgesia; Natural Childbirth
Keywords: Acupuncture; pain relief; labour; randomized controlled trial; TENS
MeSH Terms: interventions — Acupuncture Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture Group (Experimental): Acupuncture treatment during labor
  Interventions: Procedure: Acupuncture
- TENS Group (Active Comparator): Transcutaneous Electric Nerve Stimulation (TENS treatment)during labor
  Interventions: Other: TENS
- Traditional Group (Active Comparator): Traditional pain treatment during labor
  Interventions: Other: Traditional Group

INTERVENTIONS:
Procedure: Acupuncture — Based on international experiences and experiences from the pilot project 34 specified acupuncture points could be used.Treatment was individualised according to the woman's mobility and localization of pain. Needles were sterile stainless steel acupuncture needles in three lengths: 0.20 x 15 mm, 0.30 x 30 mm and 0.35 x 50 mm. No electric stimulation was used. The duration of needling could vary from 30 minutes to two hours and could be repeated. The needles were removed if the patient felt uncomfortable or in cases with obstetric pathology.
  Arms: Acupuncture Group
Other: TENS — The Transcutaneous Electric Nerve Stimulation (TENS treatment) was carried out using a B.C - TENS 120Z unit. Two to four electrodes were placed on the skin of the lower back. The units were set in constant mode, initially with a pulse width of 60 micro-seconds and a pulse rate of 100 pulses per second. The treatment lasted from 20 to 45 minutes and could be repeated. The intensity of stimulation could be adjusted by the woman or the midwife.
  Arms: TENS Group
Other: Traditional Group — All analgesic methods available (Sterile water papules, nitro oxygen, bath tub, pethidine and epidural analgesics (EDA)). A specific analgesic was chosen by the woman and the midwife after informed choice.
  Other Names: Tratitional analgesic
  Arms: Traditional Group

SUMMARY:
The purpose of this study is to investigate the effect of acupuncture for pain relief and relaxation during childbirth.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of acupuncture for pain relief an relaxation during childbirth.

In a controlled study 607 healthy patients in active labor at term are randomly assigned to receive either acupuncture, TENS or traditional analgesia. Pharmacological analgesia is provided on request. The treatment is administered by midwives trained in acupuncture and TENS. The objective parameter of outcome is the need for conventional analgesia in each group. Visual analogue scale assessments are used to evaluate participants perception of pain before, during and after treatment. Questionnaires filled out two months after delivery is used to investigate the patients experience and satisfaction with delivery and analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, Danish speaking women with a normal singleton pregnancy giving birth at term 37 - 42 weeks) with a fetus in cephalic presentation.

Exclusion Criteria:

* Women with medical diseases or complicated pregnancy. Women who has already received conventional analgesia during labor.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2001-03; Primary Completion 2004-02 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
The need for conventional analgesic in each group. | during labor

SECONDARY OUTCOMES:
Obstetric outcome: duration of labour, use of oxytocin, incidence of caesarean section, bleeding, apgar score, cord blood pH | from randomization until birth
visual analogue scale is used to evaluate subjective effect on pain. | Just before randomization, one hour after randomization and subsequently every two hours until the child was born
Questionaries filled out by the parturients to investigate satisfactory with analgesic given. | two months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lone Hvidman, MD,PhD, Study Chair — Department of Obstetrics, Aarhus University Hospital, Skejby, Denmark; Morten Hedegaard, MD, PhD, Study Chair — Department Obstetrics, Rigshospitalet, Denmark; Lissa Borup, Midwife, Principal Investigator — Department of Obstetrics, Aarhus University Hospital, Skejby; Winnie M. Wurlitzer, Midwife, Principal Investigator — Department of obstetrics, Aarhus University Hospital, Skejby
Locations (1):
- Dept Obstetrics, Aarhus University Hospital, Skejby, Aarhus, Denmark